CLINICAL TRIAL: NCT03232567
Title: Single-ascending-dose Study of the Safety and Immunogenicity of NasoVAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: ALT103-201
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Results first posted 2019-04-11 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Single ascending dose study
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NasoVAX low dose (Experimental): NasoVAX administered by intranasal spray at a single dose of 1×10(9th) viral particles (vp) versus placebo
  Interventions: Biological: NasoVAX
- NasoVAX medium dose (Experimental): NasoVAX administered by intranasal spray at a single dose of 1×10(10th) viral particles (vp) versus placebo
  Interventions: Biological: NasoVAX
- NasoVAX high dose (Experimental): NasoVAX administered by intranasal spray at a single dose of 1×10(11th) viral particles (vp) versus placebo
  Interventions: Biological: NasoVAX
- Placebo (Placebo Comparator): Normal saline administered by intranasal spray at a single dose
  Interventions: Biological: NasoVAX

INTERVENTIONS:
Biological: NasoVAX — Single ascending dose study

SUMMARY:
This is a Phase 2a, randomized, double-blind, placebo-controlled trial to evaluate the safety and immunogenicity of NasoVAX in healthy adults 18 to 49 years of age. Subjects will be screened within 28 days of randomization (Day 1).

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, double-blind, placebo-controlled trial to evaluate the safety and immunogenicity of NasoVAX in healthy adults 18 to 49 years of age. Subjects will be screened within 28 days of randomization (Day 1). Approximately 60 subjects who meet all inclusion and no exclusion criteria and provide written informed consent will be enrolled into 3 sequential cohorts of 20 subjects each defined by the viral particle dose (1×10(9th), 1×10(10th), and 1×10(11th) vp). Within each cohort and its sentinel group, subjects will be randomized in a 3:1 ratio to receive 1 intranasal dose of NasoVAX or placebo (Day 1). A sentinel group of 5 subjects from each cohort will be dosed and followed through Day 8. Dosing of the remainder of each cohort may proceed if no events meeting stopping criteria have occurred. The SRC, consisting of the Investigator, the Medical Monitor, and a Sponsor Representative, will review AE, reactogenicity, and laboratory data through Day 8 for all subjects in each cohort before subjects are randomized to the next higher dose. If any event meeting stopping criteria occur, the SRC will review all available safety information before additional patients are dosed.

ELIGIBILITY:
Subjects who meet all of the following criteria may be included in the study:

1. Men and women 18 to 49 years of age, inclusive
2. Good general health status as determined by the Investigator
3. Adequate venous access for repeated phlebotomies
4. Screening laboratory results within institutional normal range or Grade 1 elevation if the Investigator documents clinical insignificance. Creatine kinase or bilirubin may be Grade 2 if associated with normal alanine aminotransferase (ALT) and aspartate aminotransferase (AST) and the Investigator considers the result not to be clinically significant due to vigorous exercise or Gilbert's syndrome
5. Negative drug and alcohol screen at Screening and predose on Day 1
6. For women who have not been surgically sterilized or have laboratory confirmation of postmenopausal status, negative pregnancy test
7. Willingness to practice a highly effective method of contraception that may include, but is not limited to, abstinence, sex only with persons of the same sex, monogamous relationship with a postmenopausal partner, monogamous relationship with vasectomized partner, vasectomy, surgical sterilization (hysterectomy, or bilateral tubal ligation, salpingectomy, or oophorectomy), licensed hormonal methods, intrauterine device (IUD), or consistent use of a barrier method (eg, condom, diaphragm) with spermicide for 28 days after the NasoVAX/placebo dose
8. Willingness to participate and comply with all aspects of the study through the entire study period, including nasopharyngeal swabs and blood and urine samples
9. Provision of written informed consent

Subjects who meet any of the following criteria will be excluded from the study:

1. Pregnant, possibly pregnant, or lactating women
2. Household contacts of pregnant women, children < 5 years of age, or immunocompromised individuals for the period up through 2 weeks postvaccination
3. Persons who care for pregnant women, children < 5 years of age, or immunocompromised individuals for the period up through 2 weeks postvaccination
4. Body mass index > 35.0 kg/m2
5. Positive results for HIV, hepatitis B virus, or hepatitis C virus at Screening
6. Asthma or other chronic lung disease that is greater than mild in severity. Specifically excluded are participants with the any of the following events in the past year:

   * Daily symptoms
   * Daily use of short acting beta 2 agonists
   * Use of inhaled steroids or theophylline
   * Use of pulse systemic steroids
   * Emergency care or hospitalization related to asthma or other chronic lung disease
   * Systemic steroids for asthma exacerbation
7. History of diabetes mellitus (gestational diabetes is allowed if treatment was not required postpartum and serum glucose is currently in the normal range)
8. History of coronary artery disease, arrhythmia, or congestive heart failure
9. Clinically significant ECG abnormality as determined by the Investigator
10. Poorly controlled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 95 mmHg) at Screening or predose on Day 1
11. History of anaphylaxis or angioedema
12. Known allergy to any of the ingredients in the vaccine formulation
13. History of chronic rhinitis, nasal septal defect, cleft palate, nasal polyps, or other nasal abnormality that might affect vaccine administration
14. Previous nasal surgery or nasal cauterization
15. Any symptoms of upper respiratory infection or temperature > 38°C within 3 days before Day 1
16. Any symptoms within 24 hours before Day 1 of upper respiratory illness of allergy flare-up that, in the opinion of the Investigator, presents as nasal congestion or rhinorrhea that could inhibit the proper administration of the IP
17. Known or suspected malignancy, excluding non-melanoma skin cancers and other early stage surgically excised malignancies that the Investigator considers to be exceedingly unlikely to recur
18. Immunocompromised individuals, including those who have used corticosteroids (including intranasal steroids), alkylating drugs, antimetabolites, radiation, immune-modulating biologics, or other immunomodulating therapies within 90 days before Day 1 or those who plan use during the study period
19. Use of statin medication within 30 days before Day 1 (see list in Section 6.8.1)
20. Receipt of intranasal medications (including over-the-counter medications) within 30 days before Day 1
21. Receipt of any investigational product (IP) within 30 days before Day 1
22. Receipt of any vaccine within 30 days before Day 1
23. Receipt of intranasal vaccine within 90 days before Day 1
24. Receipt of any influenza vaccine within 6 months before Day 1
25. Any change in medication for a chronic medical condition within 30 days before Day 1
26. Past regular use or current use of intranasal illicit drugs
27. Smoking of any type (eg, cigarettes, electronic cigarettes, marijuana) or use of any tobacco product within 30 days before Day 1
28. Any medical, psychiatric, or social condition or occupational or other responsibility that in the judgment of the Investigator would interfere with or serve as a contraindication to protocol adherence, assessment of safety (including reactogenicity), or a subject's ability to give informed consent

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bart, MD, Principal Investigator — Optimal Research
Locations (1):
- Optimal Health Research, Rockville, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 2a, randomized, double-blind, placebo-controlled trial to evaluate the safety and immunogenicity of NasoVAX in healthy adults 18 to 49 years of age. Subjects were screened within 28 days of randomization.
Pre-assignment Details: 60 subjects who met all inclusion and no exclusion criteria and provided written informed consent were enrolled into 3 sequential cohorts of 20 subjects each defined by the vaccine dose (1×10^9, 1×10^10,1×10^11 vp). Within each cohort and its sentinel group, subjects were randomized in a 3:1 ratio to receive 1 intranasal dose of NasoVAX or placebo
Groups:
- NasoVAX Low Dose: NasoVAX administered by intranasal spray at a single dose of 1×10^9 viral particles (vp)
- NasoVAX Medium Dose: NasoVAX administered by intranasal spray at a single dose of 1×10^10 viral particles (vp)
- NasoVAX High Dose: NasoVAX administered by intranasal spray at a single dose of 1×10^11 viral particles (vp)
Period: Overall Study
Arm/Group | NasoVAX Low Dose | NasoVAX Medium Dose | NasoVAX High Dose | Placebo
Started | 15 | 15 | 15 | 15
Completed | 15 | 14 | 15 | 15
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- NasoVAX Low Dose: NasoVAX administered by intranasal spray at a single dose of 1×10^9viral particles (vp)
- Total: Total of all reporting groups
Arm/Group | NasoVAX Low Dose | NasoVAX Medium Dose | NasoVAX High Dose | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 0 | 0 | 0 | 0 | 0
  Age: Between 18 and 65 years | 15 | 15 | 15 | 15 | 60
  Age: >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 30.1 [19 to 47] | 31.6 [18 to 46] | 32.6 [21 to 48] | 29.3 [20 to 45] | 30.9 [18 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 6 | 6 | 33
  Male | 4 | 5 | 9 | 9 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 2 | 0 | 9
  Not Hispanic or Latino | 12 | 11 | 13 | 15 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 5 | 6 | 20
  White | 7 | 7 | 7 | 9 | 30
  More than one race | 1 | 2 | 1 | 0 | 4
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Emergent Adverse Events in Participants [Safety and Tolerability]
Description: Adverse events (AEs): counts and percentages of subjects with AEs Day 1 to day 29 and Medically attended AEs (MAEs), serious AEs (SAEs), new-onset chronic illnesses (NCIs) from Day 1 to Day 181
Time Frame: Day 1 to Day 181
Population: All ALT-103-201 and ALT-FLZ-401 subjects who provide informed consent, are randomized, and receive at least 1 vaccination. The Safety Population will be used for all safety analyses and will be analyzed according to the treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- NasoVAX Low Dose: NasoVAX administered by intranasal spray at a single dose of 1×10^9 viral particles (vp) versus placebo
  NasoVAX: Single ascending dose study
- NasoVAX Medium Dose: NasoVAX administered by intranasal spray at a single dose of 1×10^10 viral particles (vp) versus placebo
  NasoVAX: Single ascending dose study
- NasoVAX High Dose: NasoVAX administered by intranasal spray at a single dose of 1×10^11 viral particles (vp) versus placebo
  NasoVAX: Single ascending dose study
Arm/Group | NasoVAX Low Dose | NasoVAX Medium Dose | NasoVAX High Dose | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants
  Any TEAE | 10 | 10 | 10 | 15
  Serious TEAE | 0 | 0 | 0 | 0
  IP Related TEAE | 2 | 5 | 3 | 3
  IP Related SAE | 0 | 0 | 0 | 0
  Grade 3 or 4 TEAE | 0 | 2 | 1 | 0
  TEAE Leading to Withdrawal | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Treatment-Emergent Reactogenicity Events in Participants [Safety and Tolerability]
Description: Reactogenicity: counts and percentages of subjects with 'yes' to any reactogenicity event (nasal irritation, sneezing, nasal congestion, sore throat, change in smell, change in taste, change in vision, eye pain, headache, fatigue, muscle ache, nausea, vomiting, diarrhea, chills, fever)
Time Frame: 14-days after vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NasoVAX Low Dose | NasoVAX Medium Dose | NasoVAX High Dose | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants
  Any local event | 9 | 9 | 6 | 6
  Any systemic event | 9 | 11 | 5 | 6

3. Secondary Outcome: Geometric Mean Antibody Level Measured by Hemagglutination Inhibition (HAI) in Serum
Description: The antilog of the mean of the log-transformed antibody titers for humoral immune response to NasoVAX at Day 29 by HAI
Time Frame: Day 1 to Day 29
Population: Per-protocol population: All subjects who received the assigned dose of the test article, had HAI assay results on Days 1 and 29, and had no major protocol deviations affecting the primary immunogenicity outcomes.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | NasoVAX Low Dose | NasoVAX Medium Dose | NasoVAX High Dose | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Titer | 87.2 [52.7 to 144.3] | 136.1 [81.7 to 226.6] | 164.0 [99.0 to 271.6] | 31.3 [18.9 to 52.0]

4. Secondary Outcome: Geometric Mean Ratio of Postvaccination and Prevaccination Antibody Level Measured by Hemagglutination Inhibition (HAI) in Serum
Description: The ratio of postvaccination and prevaccination geometric mean titers within the same dose group for humoral immune response to NasoVAX at Day 29 by HAI
Time Frame: Day 1 to Day 29
Population: Per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | NasoVAX Low Dose | NasoVAX Medium Dose | NasoVAX High Dose | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Ratio | 2.1 [1.1 to 4.2] | 2.2 [1.2 to 4.3] | 4.3 [1.5 to 12.0] | 0.9 [0.7 to 1.2]

5. Secondary Outcome: Seroprotection Rate
Description: The percentage of subjects with an HAI titer greater than or equal to 1:40
Time Frame: Day 1 to Day 29
Population: Per-protocol population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NasoVAX Low Dose | NasoVAX Medium Dose | NasoVAX High Dose | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
percentage of participants | 80.0 [51.9 to 95.7] | 100 [78.2 to 100] | 100 [78.2 to 100] | 53.3 [26.6 to 78.7]
Statistical Analysis 1: Comparison: NasoVAX Low Dose vs Placebo; Test type: Superiority; p = 0.2451, Fisher Exact
Statistical Analysis 2: Comparison: NasoVAX Medium Dose vs Placebo; Test type: Superiority; p = 0.0063, Fisher Exact
Statistical Analysis 3: Comparison: NasoVAX High Dose vs Placebo; Test type: Superiority; p = 0.0063, Fisher Exact

6. Secondary Outcome: Seroconversion Rate
Description: The percentage of subjects with either a baseline HAI titer less than 1:10 and a postvaccination titer greater than or equal to 1:40 or a baseline HAI titer greater than or equal to 1:10 and a 4-fold increase in postvaccination HAI titer relative to baseline
Time Frame: Day 1 to Day 29
Population: Per-protocol population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NasoVAX Low Dose | NasoVAX Medium Dose | NasoVAX High Dose | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
percentage of participants | 13.3 [1.7 to 40.5] | 26.7 [7.8 to 55.1] | 33.3 [11.8 to 61.6] | 0.0 [0.0 to 21.8]
Statistical Analysis 1: Comparison: NasoVAX Low Dose vs Placebo; Test type: Superiority; p = 0.4828, Fisher Exact
Statistical Analysis 2: Comparison: NasoVAX Medium Dose vs Placebo; Test type: Superiority; p = 0.0996, Fisher Exact
Statistical Analysis 3: Comparison: NasoVAX High Dose vs Placebo; Test type: Superiority; p = 0.0421, Fisher Exact

7. Secondary Outcome: Antibody Level Measured by Microneutralization in Serum
Description: Geometric mean titer (GMT) for humoral immune response to NasoVAX at Day 29 by microneutralization
Time Frame: Day 1 to Day 29
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | NasoVAX Low Dose | NasoVAX Medium Dose | NasoVAX High Dose | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Titer | 44.9 [21.8 to 92.3] | 113.1 [58.0 to 220.8] | 142.5 [93.6 to 217.1] | 17.8 [9.1 to 35.0]

8. Secondary Outcome: Antibody Responder Rate by Microneutralization
Description: The percentages of subjects with 2-fold and 4-fold rises from baseline in antibody level measured by microneutralization
Time Frame: Day 1 to Day 29
Population: Per-protocol population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NasoVAX Low Dose | NasoVAX Medium Dose | NasoVAX High Dose | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
percentage of participants
  Percentage of subjects with 2-fold rise | 40.0 [16.3 to 67.7] | 46.7 [21.3 to 73.4] | 73.3 [44.9 to 92.2] | 0.0 [0.0 to 21.8]
  Percentage of subjects with 4-fold rise | 13.3 [1.7 to 40.5] | 26.7 [7.8 to 55.1] | 53.3 [26.6 to 78.7] | 0.0 [0.0 to 21.8]
Statistical Analysis 1: Comparison: NasoVAX Low Dose vs Placebo; NasoVAX low dose vs placebo; Test type: Superiority; p = 0.0169, Fisher Exact
Statistical Analysis 2: Comparison: NasoVAX Medium Dose vs Placebo; NasoVAX medium dose vs placebo; Test type: Superiority; p = 0.0063, Fisher Exact
Statistical Analysis 3: Comparison: NasoVAX High Dose vs Placebo; NasoVAX high dose vs placebo; Test type: Superiority; p < 0.0001, Fisher Exact

ADVERSE EVENTS:
Time Frame: AEs Day 1 to day 29 Medically attended AEs (MAEs), serious AEs (SAEs), new-onset chronic illnesses (NCIs) from Day 1 to Day 181
Description: Adverse events (AEs): counts and percentages of subjects with AEs Day 1 to day 29 and Medically attended AEs (MAEs), serious AEs (SAEs), new-onset chronic illnesses (NCIs) from Day 1 to Day 181
Groups:
- Placebo: Normal saline administered
Arm/Group | NasoVAX Low Dose | NasoVAX Medium Dose | NasoVAX High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 10/15 | 10/15 | 10/15 | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NasoVAX Low Dose (N=15) | NasoVAX Medium Dose (N=15) | NasoVAX High Dose (N=15) | Placebo (N=15)
Any treatment emergent adverse event (Product Issues) | 10 | 10 | 10 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT03232567/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT03232567/SAP_001.pdf